CLINICAL TRIAL: NCT03518073
Title: Assessment of Safety, Tolerability, and Efficacy of LY3303560 in Early Symptomatic Alzheimer's Disease
Brief Title: A Study of LY3303560 in Participants With Early Symptomatic Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16124; I8G-MC-LMDC (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease (AD)
Keywords: Memory problems; Cognitive impairment; PERISCOPE-ALZ; Dementia; Tauopathy; Neurofibrillary tangles
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders; Cognitive Dysfunction; Dementia; Tauopathies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received intravenous (IV) infusion of placebo once every four weeks (Q4W) for 100 weeks.
  Interventions: Drug: Placebo
- Zagotenemab 1400 mg (Experimental): Participants received IV infusion of 1400 milligram (mg) zagotenemab Q4W for 100 weeks.
  Interventions: Drug: Zagotenemab
- Zagotenemab 5600 mg (Experimental): Participants received IV infusion of 5600 mg zagotenemab Q4W for 100 weeks.
  Interventions: Drug: Zagotenemab

INTERVENTIONS:
Drug: Zagotenemab — Administered IV
  Other Names: LY3303560
  Arms: Zagotenemab 1400 mg; Zagotenemab 5600 mg
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a study drug that targets an abnormal protein in the brain found in people with Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have gradual and progressive change in memory function for >6 months.
* Participants must have a family member or close friend who is with you at least 10 hours per week and can attend study appointments.

Exclusion Criteria:

* Participants must not have significant neurological disease affecting the nervous system, other than AD, that affects cognition or may affect completion of the study.
* Participants must not have serious or unstable illness that could interfere with the analysis of the study or has a life expectancy <24 months.
* Participants must not have history of cancer within the last 5 years with the exception of certain types of skin, cervical, prostate, and other cancers that are not likely to recur or spread.
* Participants must not have serious risk for suicide.
* Participants must not have history of drug or alcohol use disorder within the last 2 years.
* Participants must not have multiple severe drug allergies
* Participants must not have HIV, Hepatitis B or Hepatitis C
* Participants must not be receiving gamma globulin (IgG) or intravenous immunoglobulin (IVIG) therapy

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (60):
- United States (49):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Pharmacology Research Institute, Encino, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Irvine Clinical Research Center, Irvine, California
  - Pharmacology Research Institute, Los Alamitos, California
  - National Research Institute - Huntington Park, Panorama City, California
  - Anderson Clinical Research, Redlands, California
  - Pacific Research Network, San Diego, California
  - Univ of California San Francisco, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - New England Institute for Clinical Research, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Julie B. Schwartzbard, MD, PA, Aventura, Florida
  - Quantum Laboratories Clinical Research, Deerfield Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - VIN-Victor Faradji, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - BioClinica Inc, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Brain Matters Research, Stuart, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Columbus Memory Center, PC, Columbus, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - AMITA Health - Alexian Brothers Neurosciences Institute Clinical Research, Elk Grove Village, Illinois
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Rowe Neurology Institute, Lenexa, Kansas
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Clinical Research Professionals, Chesterfield, Missouri
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Lindner Research Center, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Cincinnati Health Neurology, Dayton, Ohio
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Baylor AT&T Memory Center, Dallas, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Houston Methodist Research Ins, Houston, Texas
  - The Memory Clinic, Bennington, Vermont
  - Cognition Health, Fairfax, Virginia
- Canada (5):
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ca-on
  - Toronto Memory Program, Toronto, Ontario
  - Clinique de la Mémoire de l'Outaouais, Gatineau, Quebec
  - NeuroSearch Developements, Greenfield Park, Quebec
  - Q&T Research Sherbrooke Inc., Sherbrooke, Quebec
- Japan (6):
  - National Center for Geriatrics and Gerontology, Ōbu, Aichi-ken
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Nippon Medical School Hospital, Tokyo, Jp-13
  - National hospital Organization Utano National Hospital, Kyoto, Jp-26
  - Katayama Medical Clinic, Kurashiki, Jp-33
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Fleisher AS, Munsie LM, Perahia DGS, Andersen SW, Higgins IA, Hauck PM, Lo AC, Sims JR, Brys M, Mintun M; PERISCOPE-ALZ Site Investigators. Assessment of Efficacy and Safety of Zagotenemab: Results From PERISCOPE-ALZ, a Phase 2 Study in Early Symptomatic Alzheimer Disease. Neurology. 2024 Mar 12;102(5):e208061. doi: 10.1212/WNL.0000000000208061. Epub 2024 Feb 22. PMID 38386949
- See also: A Study of LY3303560 in Participants With Early Symptomatic Alzheimer's Disease — https://trials.lillytrialguide.com/en-US/trial/3iXXmw7cgM8KieSEmiIuSk

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Started | 118 | 126 | 116
Received at Least One Dose of Study Drug | 118 | 126 | 116
Completed | 74 | 78 | 70
Not Completed | 44 | 48 | 46
Not completed — Adverse Event | 2 | 4 | 2
Not completed — Death | 2 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Physician Decision | 5 | 0 | 2
Not completed — Progressive disease | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 30 | 34 | 29
Not completed — Withdrawal Due To Caregiver Circumstances | 1 | 6 | 7
Not completed — Covid-19 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants received IV infusion of placebo Q4W for 100 weeks.
- Zagotenemab 1400 mg: Participants received IV infusion of 1400 mg zagotenemab Q4W for 100 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg | Total
Number analyzed (Participants) | 118 | 126 | 116 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.30 (5.22) | 75.10 (5.33) | 75.70 (5.49) | 75.40 (5.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 72 | 65 | 190
  Male | 65 | 54 | 51 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 10
  Not Hispanic or Latino | 112 | 120 | 110 | 342
  Unknown or Not Reported | 2 | 3 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 18 | 18 | 17 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 2 | 2 | 6
  White | 98 | 106 | 96 | 300
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 15 | 15 | 13 | 43
  Japan | 15 | 17 | 17 | 49
  United States | 88 | 94 | 86 | 268
Integrated Alzheimer's Disease Rating Scale (iADRS) [Mean (Standard Deviation); unit: score on a scale] — Integrated Alzheimer's Disease Rating Scale (iADRS) is a simple linear combination of scores from 13-item alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). It is used to assess whether zagotenemab slows down the cognitive and functional decline associated with early symptomatic Alzheimer's Disease, compared to placebo. The iADRS score ranges from 0 to 144 with lower scores indicating worse performance and higher score better performance. Population: All randomized participants with iADRS data at baseline.
  score on a scale
    number analyzed (Participants) | 118 | 124 | 114 | 356
    (all) | 103.50 (13.51) | 105.96 (13.34) | 103.60 (11.65) | 104.39 (12.90)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS)
Description: Integrated Alzheimer's Disease Rating Scale (iADRS) is a simple linear combination of scores from 13-item alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). It is used to assess whether zagotenemab slows down the cognitive and functional decline associated with early symptomatic Alzheimer's Disease, compared to placebo. The iADRS score ranges from 0 to 144 with lower scores indicating worse performance and higher score better performance. Change from baseline was calculated using Bayesian disease progression model (DPM) with fixed, categorical effects of treatment, pooled site, acetylcholinesterase inhibitor (AChEI) use at baseline (yes/no), and the continuous effects of baseline score and age at baseline. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 104
Population: All randomized participants with baseline, post-baseline iADRS data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 70 | 72 | 68
score on a scale | -13.72 [-15.325 to -12.161] | -15.11 [-16.779 to -13.479] | -14.38 [-16.054 to -12.727]
Statistical Analysis 1: Comparison: Placebo vs Zagotenemab 1400 mg; Test type: Superiority; Posterior Mean Ratio = 1.10, 95% CI 2-sided [0.959 to 1.265] — Posterior mean ratio with 95% credible interval is reported
Statistical Analysis 2: Comparison: Placebo vs Zagotenemab 5600 mg; Test type: Superiority; Posterior Mean Ratio = 1.05, 95% CI 2-sided [0.907 to 1.209] — Posterior mean ratio with 95% credible interval is reported

2. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Assessment Scale- Cognitive Subscale (ADAS-Cog13) Score
Description: The ADAS is a rater-administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with Alzheimer's Disease (AD). The cognitive subscale of the ADAS consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation, and maze completion measures. The ADAS-Cog13 scale ranges from 0 to 85, with higher scores indicating greater disease severity. Change from baseline was calculated using Bayesian disease progression model (DPM) with fixed, categorical effects of treatment, pooled site, acetylcholinesterase inhibitor (AChEI) use at baseline (yes/no), and the continuous effects of baseline score and age at baseline. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 104
Population: All randomized participants with baseline, post-baseline ADAS-Cog13 data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 71 | 76 | 69
score on a scale | 7.13 [6.176 to 8.104] | 7.85 [6.867 to 8.848] | 6.30 [5.353 to 7.262]
Statistical Analysis 1: Comparison: Placebo vs Zagotenemab 1400 mg; Test type: Superiority; Posterior Mean Ratio = 1.11, 95% CI 2-sided [0.943 to 1.290] — Posterior mean ratio with 95% credible interval is reported
Statistical Analysis 2: Comparison: Placebo vs Zagotenemab 5600 mg; Test type: Superiority; Posterior Mean Ratio = 0.89, 95% CI 2-sided [0.737 to 1.053] — Posterior mean ratio with 95% credible interval is reported

3. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living Scale (ADCS-iADL) Score
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures basic, instrumental activities of daily living by participants (instrumental activity items 6a, 7-23). The range for the ADCS-iADL is 0-59, with lower scores indicating greater disease severity. Change from baseline was calculated using Bayesian disease progression model (DPM) with fixed, categorical effects of treatment, pooled site, acetylcholinesterase inhibitor (AChEI) use at baseline (yes/no), and the continuous effects of baseline score and age at baseline. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 104
Population: All randomized participants with baseline, post-baseline ADCS-iADL data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 72 | 74 | 69
score on a scale | -6.67 [-7.730 to -5.643] | -7.06 [-8.148 to -6.004] | -8.05 [-9.203 to -6.922]
Statistical Analysis 1: Comparison: Placebo vs Zagotenemab 1400 mg; Test type: Superiority; Posterior Mean Ratio = 1.06, 95% CI 2-sided [0.873 to 1.284] — Posterior mean ratio with 95% credible interval is reported
Statistical Analysis 2: Comparison: Placebo vs Zagotenemab 5600 mg; Test type: Superiority; Posterior Mean Ratio = 1.21, 95% CI 2-sided [1.006 to 1.453] — Posterior mean ratio with 95% credible interval is reported

4. Secondary Outcome: Change From Baseline on the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) Score
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning: memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. Change from baseline was calculated using Bayesian disease progression model (DPM) with fixed, categorical effects of treatment, pooled site, acetylcholinesterase inhibitor (AChEI) use at baseline (yes/no), and the continuous effects of baseline score and age at baseline. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 104
Population: All randomized participants with baseline, post-baseline CDR-SB data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 72 | 75 | 68
score on a scale | 2.26 [1.976 to 2.544] | 2.52 [2.233 to 2.815] | 2.14 [1.854 to 2.439]
Statistical Analysis 1: Comparison: Placebo vs Zagotenemab 1400 mg; Test type: Superiority; Posterior Mean Ratio = 1.12, 95% CI 2-sided [0.963 to 1.300] — Posterior mean ratio with 95% credible interval is reported
Statistical Analysis 2: Comparison: Placebo vs Zagotenemab 5600 mg; Test type: Superiority; Posterior Mean Ratio = 0.95, 95% CI 2-sided [0.805 to 1.119] — Posterior mean ratio with 95% credible interval is reported

5. Secondary Outcome: Change From Baseline on the Mini Mental Status Examination (MMSE) Score
Description: The MMSE is a brief instrument used to assess cognitive function. The instrument is divided into 2 sections. The first section measures orientation, memory, and attention. The maximum score for the first section is 21. The second section tests the ability of the person to name objects, follow verbal and written commands, write a sentence, and copy figures. The maximum score for the second section is 9. The range for the total MMSE score is 0 to 30, with lower scores indicating greater level of impairment. Change from baseline was calculated using Bayesian disease progression model (DPM) with fixed, categorical effects of treatment, pooled site, acetylcholinesterase inhibitor (AChEI) use at baseline (yes/no), and the continuous effects of baseline score and age at baseline. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 104
Population: All randomized participants with baseline, post-baseline MMSE data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 72 | 76 | 68
score on a scale | -4.29 [-4.858 to -3.739] | -4.44 [-4.994 to -3.901] | -3.83 [-4.40 to -3.265]
Statistical Analysis 1: Comparison: Placebo vs Zagotenemab 1400 mg; Test type: Superiority; Posterior Mean Ratio = 1.04, 95% CI 2-sided [0.880 to 1.221] — Posterior mean ratio with 95% credible interval is reported
Statistical Analysis 2: Comparison: Placebo vs Zagotenemab 5600 mg; Test type: Superiority; Posterior Mean Ratio = 0.89, 95% CI 2-sided [0.742 to 1.065] — Posterior mean ratio with 95% credible interval is reported

6. Secondary Outcome: Change From Baseline in Brain Aggregated Tau Deposition as Measured by Flortaucipir F-18 Positron Emission Tomography (PET) Scan.
Description: Deposition of abnormal tau protein in the brain associated with AD was assessed by quantitative PET scan using flortaucipir F-18. Flortaucipir is an F-18-labeled small molecule that binds with high affinity and selectivity to aggregated tau, and provides a measure of aggregated tau deposition in the brain, expressed as flortaucipir standardized uptake value ratio (SUVr). Change from baseline was calculated using mixed model repeated measures (MMRM) with fixed, categorical effects of treatment, visit, treatment-by-visit interaction, and continuous effect of baseline SUVr and age. A positive change from baseline indicates increased aggregated tau deposition that is believed to be associated with a more rapid rate of cognitive deterioration.
Time Frame: Baseline, Week 104
Population: All randomized participants with baseline, post-baseline PET tau data.
Measure: Least Squares Mean (Standard Error); unit: standardized uptake value ratio (SUVr)
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 62 | 66 | 63
standardized uptake value ratio (SUVr) | 0.08 (0.012) | 0.10 (0.011) | 0.10 (0.012)
Statistical Analysis 1: Comparison: Placebo vs Zagotenemab 1400 mg; Test type: Superiority; p = 0.253, Mixed Models Analysis; LS Mean Difference = 0.02, 95% CI 2-sided [-0.01 to 0.05], Standard Error of Mean 0.016
Statistical Analysis 2: Comparison: Placebo vs Zagotenemab 5600 mg; Test type: Superiority; p = 0.354, Mixed Models Analysis; LS Mean Difference = 0.02, 95% CI 2-sided [-0.02 to 0.05], Standard Error of Mean 0.016

7. Secondary Outcome: Change From Baseline in Brain Volume as Measured by Volumetric Magnetic Resonance Imaging (vMRI)
Description: Alzheimer's disease is also associated with pronounced brain atrophy, reflecting bulk neurodegenerative loss of gray and white matter. Progression of brain atrophy is assessed by vMRI, providing regional quantification of volume loss. Negative change from baseline indicates greater disease severity. Change from baseline was calculated using mixed model repeated measures (MMRM) with fixed, categorical effects of treatment, visit, treatment-by-visit interaction, and continuous effect of baseline vMRI, baseline intracranial volume (ICV) and age.
Time Frame: Baseline, Week 104
Population: All randomized participants with baseline, post-baseline vMRI brain volume data.
Measure: Least Squares Mean (Standard Error); unit: cubic centimeter (cm^3)
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 64 | 65 | 57
cubic centimeter (cm^3) | -24.06 (1.101) | -23.44 (1.095) | -23.55 (1.158)
Statistical Analysis 1: Comparison: Placebo vs Zagotenemab 1400 mg; Test type: Superiority; p = 0.691, Mixed Models Analysis; LS Mean Difference = 0.62, 95% CI 2-sided [-2.44 to 3.68], Standard Error of Mean 1.554
Statistical Analysis 2: Comparison: Placebo vs Zagotenemab 5600 mg; Test type: Superiority; p = 0.749, Mixed Models Analysis; LS Mean Difference = 0.51, 95% CI 2-sided [-2.64 to 3.66], Standard Error of Mean 1.599

8. Secondary Outcome: Number of Participants With Suicidal Ideation and Behaviors Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviours, and has a binary response (yes/no).
  * Suicidal Ideation: a "yes" answer to any one of 5 suicidal ideation questions: Wish to be Dead, Non-specific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Active Suicidal Ideation with Some Intent to Act without Specific Plan, Active Suicidal Ideation with Specific Plan and Intent.
  * Suicidal Behaviour: a "yes" answer to any of 5 suicidal behaviour questions: Preparatory Acts or Behaviour, Aborted Attempt, Interrupted Attempt, Actual Attempt (non-fatal), Completed Suicide.
Time Frame: Baseline through Week 104
Population: All randomized participants who received at least one dose of study drug and had baseline, at least one post baseline C-SSRS assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 118 | 126 | 116
Participants
  Suicidal Ideation | 5 | 5 | 5
  Suicidal Behaviour | 1 | 2 | 0

9. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Drug Antibodies (TE-ADA) to Zagotenemab
Description: A TE-ADA evaluable subject is considered to be TE-ADA positive:
  * If the subject has at least one post baseline titer that is a 4-fold or greater increase in titer from baseline measurement (treatment-boosted).
  * If baseline result is ADA Not Present, then the subject is TE ADA positive if there is at least one postbaseline result of ADA Present with titer >= 1:10 (treatment-induced).
Time Frame: Baseline through Week 113
Population: All randomized participants who received at least one dose of zagotenemab and had baseline, at least one post baseline ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Zagotenemab 1400 mg | Zagotenemab 5600 mg
Number analyzed (Participants) | 126 | 115
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline through End of Study (Up To 113 Weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | Zagotenemab 1400 mg | Zagotenemab 5600 mg
All-Cause Mortality (participants affected / at risk) | 2/118 | 1/126 | 3/116
Serious Adverse Events (participants affected / at risk) | 14/118 | 22/126 | 19/116
Other Adverse Events (participants affected / at risk) | 61/118 | 68/126 | 71/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=118) | Zagotenemab 1400 mg (N=126) | Zagotenemab 5600 mg (N=116)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/53 (0) | 0/72 (0) | 1/65 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/65 (1) | 0/54 (0) | 0/51 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (4) | 2 (2) | 1 (2)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Infarction (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=118) | Zagotenemab 1400 mg (N=126) | Zagotenemab 5600 mg (N=116)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 10 (12) | 11 (13)
Nausea (Gastrointestinal disorders) | 2 (3) | 7 (10) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (8) | 5 (10)
Fatigue (General disorders) | 4 (4) | 5 (5) | 6 (7)
Gait disturbance (General disorders) | 0 (0) | 7 (7) | 4 (4)
Nasopharyngitis (Infections and infestations) | 12 (13) | 5 (5) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 8 (10) | 4 (4) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 16 (28) | 18 (23) | 15 (18)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 7 (8)
Skin laceration (Injury, poisoning and procedural complications) | 7 (11) | 9 (9) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 10 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 9 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5) | 8 (8)
Dizziness (Nervous system disorders) | 10 (13) | 10 (16) | 11 (16)
Headache (Nervous system disorders) | 7 (7) | 5 (9) | 6 (7)
Anxiety (Psychiatric disorders) | 7 (9) | 4 (5) | 9 (11)
Depression (Psychiatric disorders) | 2 (2) | 5 (6) | 6 (6)
Insomnia (Psychiatric disorders) | 4 (4) | 7 (7) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (6) | 7 (7)
Hypertension (Vascular disorders) | 3 (3) | 7 (7) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03518073/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03518073/SAP_001.pdf